CLINICAL TRIAL: NCT04714372
Title: Study of FT538 in Combination With Daratumumab in Acute Myeloid Leukemia
Brief Title: FT538 in Combination With Daratumumab in AML Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2020LS114; MT2020-33 (Other: University of Minnesota Masonic Cancer Center)
Record Dates: First submitted 2021-01-14; First posted 2021-01-19 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Acute Myeloid Leukemia; Myeloid Leukemia; Monocytic Leukemia
Keywords: FT538, AML, Daratumumab, CD38
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid; Leukemia, Monocytic, Acute | interventions — daratumumab; fludarabine; fludarabine phosphate; Cyclophosphamide

STUDY DESIGN:
Intervention Model Description: This study is performed in two stages, with Stage 1 having two potential steps. A minimum of 28 days separates each patient cohort. Stage 1 step 1 uses a fast-track design (1 patient per cohort) starting at Dose Level 1. The study moves to Stage 1 Step 2 when a pre-defined adverse event occurs during fast-track enrollment, specifically, any Grade 3 non-hematologic event within 72 hours after an FT538 infusion. The cohort size increases from 1 to 3 patients with 2 additional patients added to the current cohort if the event being a Dose Limiting Toxicity (DLT) event. No intra-cohort staggering is required. Escalation in Step 2 continues until the 1st DLT event at which point Stage 2 (CRM) is activated. Stage 2 follows Continual Reassessment Method (CRM) and is initiated at the 1st DLT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Level 1: FT538 at 1 x10^8 cells/dose (Experimental): FT538 administered at assigned dose as an IV infusion via gravity on Day 1, Day 8, and Day 15
  Interventions: Drug: Daratumumab/rHuPH20; Drug: FT538; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 2: FT538 at 3 x10^8 cells/dose (Experimental): FT538 administered at assigned dose as an IV infusion via gravity on Day 1, Day 8, and Day 15
  Interventions: Drug: Daratumumab/rHuPH20; Drug: FT538; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 3: FT538 at 1 x10^9 cells/dose (Experimental): FT538 administered at assigned dose as an IV infusion via gravity on Day 1, Day 8, and Day 15
  Interventions: Drug: Daratumumab/rHuPH20; Drug: FT538; Drug: Fludarabine; Drug: Cyclophosphamide
- Dose Level 4: FT538 at 1.5 x10^9 cells/dose (Experimental): FT538 administered at assigned dose as an IV infusion via gravity on Day 1, Day 8, and Day 15
  Interventions: Drug: Daratumumab/rHuPH20; Drug: FT538; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Daratumumab/rHuPH20 — Daratumumab 1800 mg co-formulated with 30,000 units of hyaluronidase (rHuPH20) given subcutaneously into subcutaneous tissue of the abdomen approximately 3 inches [7.5 cm] to the right or left of the navel over approximately 3-5 minutes on Day -12 and Day -5 prior to the 1st FT538 infusion, and on Day +3, Day+10, and Day+17 approximately 48 hours after each FT538 infusion.
  Other Names: Darzalex
Drug: FT538 — FT538 is administered as an IV infusion via gravity using an IV administration set with an in-line filter at the patient's assigned dose levels (DL) on Day 1, Day 8, and Day 15
Drug: Fludarabine — Fludarabine 25 mg/m^2 is administered as a 1 hour intravenous (IV) infusion per institutional guidelines once a day on 2 consecutive days (Day -4, and Day -3).
  Other Names: FLUDARA
Drug: Cyclophosphamide — Cyclophosphamide 300 mg/m^2 is administered as a 2 hour intravenous (IV) infusion per institutional guidelines once a day on the same days that fludarabine is given.
  Other Names: CYTOXAN; NEOSAR

SUMMARY:
This Phase I open-label dose escalation study is conducted in two stages with a primary endpoint to identify the maximum tolerated dose (MTD) of FT538 when administered with daratumumab in patients 12 years and older with advanced acute myeloid leukemia (AML) and related myeloid diseases.

DETAILED DESCRIPTION:
FT538 is an off the shelf product comprised of allogeneic natural killer (NK)-cell immunotherapy lacking CD38 and expressing hnCD16 and IL-15RF. Daratumumab is a targeted therapy (IgG1k human monoclonal antibody) that targets CD38.

FT538 is administered once a week for 3 consecutive weeks (Day 1, Day 8, and Day 15). Up to 5 dose levels will be tested. Fixed dose subcutaneous daratumumab is given on Day -12 and Day 5 prior to the NK cells as lymphodepletion, and on Day +3, Day +10, and Day +17 to maximize targeting. A short course of outpatient lymphodepleting chemotherapy is given on Day -4 and Day -3 to promote adoptive transfer. Day 1, the day of the 1st FT538 infusion, must be a Monday.

The primary analysis for Phase I is intent-to-treat in that all patients receiving the 1st infusion of FT538 are evaluable for toxicity and efficacy. Patients who discontinue therapy prior to the first FT538 will be replaced.

There are five potential FT538 dose cohorts. The starting dose is FT538 1x10e8 cells per dose with a lower safety dose of 5x10e7 if needed (Dose Level -1). The subsequent planned FT538 cohorts are 3x10e8, 1x10e9, and 1.5 x10e9 FT538 cells per dose. Dosing is based on hnCD16 expression, where 90% ± 10% of administered FT538 cells express hnCD16. The trial is conducted with no intra-patient escalation.

ELIGIBILITY:
Disease specific Inclusion Criteria:

Acute myeloid leukemia relapsed/refractory after 2 lines of therapy; with CD38 expression

* CD38 expression is defined by ≥20% of malignant cells with CD38 expression by flow cytometry on the most recent marrow biopsy (within 30 days of enrollment - archived or fresh).
* Relapsed/refractory is defined as failure to achieve at least a Morphological Leukemia Free State (MLFS) or reverting from MLFS.
* Lines of therapy are defined as (must have had 2 prior therapies):

  * One cycle of Intensive induction chemotherapy such as 7+3, 5+2, MEC, FLAG, FLAG-Ida, CLAG ± small molecule inhibitor
  * Four weeks of HMA-based induction ± small molecule inhibitor
  * Hematopoietic stem cell transplantation (HSCT) if relapse that occurs > 90 days after HSCT
  * Gemtuzumab Ozogamicin
  * LDAC + glasdegib
  * Biomarker-specific targeted agents (FLT3 inhibitors, IDH1/2 inhibitors, others if available)
  * Other treatments could be considered after discussion with the PI

Inclusion Criteria:

* Age 12 years or older at the time of consent - Please note, enrollment of minors will be begin until permission to proceed is received from the FDA. At that time, the protocol will be updated to open enrollment to minors.
* Weight ≥ 50 kg due to FT538 fixed cell dosing and FT538 product pre-dose packaging
* Karnofsky performance status of 80-100% for 16 years and older or Lansky Play Score of 80-100 for ≥12 and < 16 years of age
* Evidence of adequate organ function within 14 days of starting study treatment defined as:

  * Estimated Glomerular Filtration Rate (estimated creatinine clearance) ≥50 mL/min/1.73m^2
  * Total bilirubin ≤ 5 × upper limit normal (ULN), not applicable for patients with Gilbert's syndrome
  * AST ≤3 × ULN and ALT ≤ 3 × ULN, not applicable if determined to be directly due to underlying malignancy
  * LVEF ≥ 40% by echocardiogram or MUGA
* Contraceptive use by men or women

  * Female subjects: Women of childbearing potential (WOCBP) must use a highly effective form of contraception from the screening visit until at least 12 months after the final dose of cyclophosphamide (CY), at least 4 months after the final dose of FT538, and at least 3 months after the final dose of daratumumab, whichever is latest.
  * Male subjects: Males with a female partner of childbearing potential or a pregnant female partner must be sterile (biologically or surgically) or use a highly effective method of contraception from the screening visit until at least 4 months after the final dose of CY and at least 4 months after the final dose of FT538, and at least 3 months after the final dose of daratumumab, whichever is latest.
* Must agree to and sign the consent for the companion Long-Term Follow-Up study (UMN CPRC #2020LS166) to fulfill the FDA required 15 years of follow-up for a genetically modified cell product.
* Must agree to and sign the consent for the companion Long-Term Follow-Up study (UMN CPRC #2020LS166) to fulfill the FDA required 15 years of follow-up for a genetically modified cell product.

Exclusion Criteria:

* Diagnosis of acute promyelocytic leukemia (APL)
* Pregnant or breastfeeding, Menstruating females of child-bearing potential must have a negative pregnancy test within 14 days of study treatment start
* Known allergy to any of study drugs or their components
* Clinically significant cardiovascular disease including any of the following: myocardial infarction within 6 months prior to first study treatment; unstable angina or congestive heart failure of New York Heart Association Grade 2 or higher or cardiac ejection fraction <40%
* Any known condition that requires systemic immunosuppressive therapy (> 5mg prednisone daily or equivalent) during the FT538 dosing period (3 days before the 1st dose through 14 days after the last dose) excluding pre-medications - inhaled and topical steroids are permitted
* Receipt of any biological therapy, chemotherapy, or radiation therapy, except for palliative purposes, within 2 weeks prior to Day 1 or five half-lives, whichever is shorter; or any investigational therapy within 28 days prior to the to the first dose of daratumumab. Maintenance hydroxyurea for blast control up to the initiation of lympho-conditioning is permitted
* Known active central nervous system (CNS) involvement or treated CNS disease that has not cleared. If prior disease related CNS involvement must have completed effective treatment of their CNS disease at least 2 months prior to Day 1 with no evidence of disease clinically and at least stable findings on relevant CNS imaging
* Non-malignant CNS disease such as epilepsy, CNS vasculitis, or neurodegenerative disease or receipt of medications for these conditions in the 2-year period leading up to study enrollment
* Clinically significant untreated/uncontrolled infection
* Live vaccine <6 weeks prior to start of lympho-conditioning
* Known seropositive for HIV or known active Hepatitis B or C infection with detectable viral load by PCR
* Prior solid organ transplant
* Allogeneic HSCT relapse occurring <90 days after HSCT
* Active graft-versus-host-disease (GvHD) requiring systemic immunosuppression within 14 days prior to enrollment
* Presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to the participant.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Maakaron, MD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose
Started | 1 | 1 | 1 | 6
Completed | 1 | 1 | 1 | 2
Not Completed | 0 | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose | Total
Number analyzed (Participants) | 1 | 1 | 1 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 1 | 4 | 6
  >=65 years | 1 | 0 | 0 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 6 | 8
  Male | 0 | 0 | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 1 | 6 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1
  White | 1 | 1 | 0 | 6 | 8
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose Limiting Toxicity (DLT) Events
Description: Dose limiting toxicity (DLT) is defined as any AE (based on CTCAE v5) that is at least possibly related to FT538 that occurs after the first FT538 infusion through the end of the DLT assessment period on Day 29 as defined below:
  Any Grade 4 non-hematologic AE, Grade 3 pulmonary or cardiac AE of any duration, Grade 3 immune cell associated neurotoxicity syndrome (ICANS) of any duration, Any other Grade 3 non-hematologic AE of >72 hours duration or Grade ≥2 acute GvHD requiring systemic steroid administration
Time Frame: 42 days from the 1st FT538 infusion
Measure: Number (90% Confidence Interval); unit: Count of Participants
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose
Number analyzed (Participants) | 1 | 1 | 1 | 6
Count of Participants | 0 [0 to 0.89] | 0 [0 to 0.89] | 0 [0 to 0.89] | 0 [0 to 0.31]

2. Secondary Outcome: Number of Participants Achieving Complete Remission (CR + CRi)
Description: Efficacy of treatment is measured by the objective response rate (Complete Remission [CR] + Complete Remission with Incomplete Hematologic Recovery [CRi]) assessed by Day 28 based on the 2017 European LeukemiaNet (ELN) response criteria CR - defined as bone marrow blast <5%, absence of circulating blasts and blasts with auer rods, absence of extramedullary disease, Absolute neutrophil count >= 1.0 × 10e9/L (1000/μL) and platelet count >=100 × 10e9/L 100,000/μL) CRi - defined as all CR criterial except for residual neutropenia (<1.0 × 10e9/L [1000/μL]) or thrombocytopenia (<100 × 10e9/L [100,000/μL])
Time Frame: 28 days from the 1st FT538 infusion
Measure: Number (90% Confidence Interval); unit: Count of Participants
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose
Number analyzed (Participants) | 1 | 1 | 1 | 6
Count of Participants | 0 [0 to 0.89] | 0 [0 to 0.89] | 0 [0 to 0.89] | 2 [0.72 to 3.9]

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as number of patients who have a partial or complete response to therapy divided by the total number of patients who received treatment.
  Response criteria will be based on 2017 European LeukemiaNet (ELN) response criteria assessing the bone marrow blast percentage, presence/absence of circulating blasts, presence/absence of blasts with auer rods, presence/absence of extramedullary disease, Absolute neutrophil counts per liter pf blood and platelet counts per liter blood
Time Frame: 12 months from the 1st FT538 infusion
Measure: Number (90% Confidence Interval); unit: participants
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose
Number analyzed (Participants) | 1 | 1 | 1 | 6
participants | 0 [0 to 0.89] | 0 [0 to 0.89] | 0 [0 to 0.89] | 2 [0.72 to 3.9]

4. Secondary Outcome: Percentage of Participants With Progression Free Survival (PFS)
Description: Percentage of participants experiencing progression free survival at one year follow up
Time Frame: 12 months from the 1st FT538 infusion
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose
Number analyzed (Participants) | 1 | 1 | 1 | 6
Percentage of participants | 0 [0 to 0.89] | 100 [0.10 to 100] | 0 [0 to 0.89] | 33 [12 to 65]

5. Secondary Outcome: Percentage of Participants With Overall Survival (OS)
Description: Percentage of participants with Overall Survival (OS) at one year follow up
Time Frame: 12 months from the 1st FT538 infusion
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose
Number analyzed (Participants) | 1 | 1 | 1 | 6
Percentage of participants | 0 [0 to 0.89] | 100 [0.10 to 100] | 0 [0 to 0.89] | 33 [12 to 65]

6. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: Number of participants experiencing adverse events with the combination of Daratumumab and FT538
Time Frame: 12 months from the 1st FT538 infusion
Measure: Number; unit: Count of Participants
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose
Number analyzed (Participants) | 1 | 1 | 1 | 6
Count of Participants | 1 | 1 | 1 | 6

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Dose Level 1: FT538 at 1 x10^8 Cells/Dose | Dose Level 2: FT538 at 3 x10^8 Cells/Dose | Dose Level 3: FT538 at 1 x10^9 Cells/Dose | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose
All-Cause Mortality (participants affected / at risk) | 1/1 | 0/1 | 1/1 | 4/6
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 5/6
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 1/1 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: FT538 at 1 x10^8 Cells/Dose (N=1) | Dose Level 2: FT538 at 3 x10^8 Cells/Dose (N=1) | Dose Level 3: FT538 at 1 x10^9 Cells/Dose (N=1) | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose (N=6)
Other, specify - Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Choledocolithiasis (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Febrile neutropenia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Level 1: FT538 at 1 x10^8 Cells/Dose (N=1) | Dose Level 2: FT538 at 3 x10^8 Cells/Dose (N=1) | Dose Level 3: FT538 at 1 x10^9 Cells/Dose (N=1) | Dose Level 4: FT538 at 1.5 x10^9 Cells/Dose (N=6)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 1 (3) | 0 (0) | 3 (3)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 4 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 4 (4)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (6)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (2) | 2 (3)
Fever (General disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Generalized edema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Viremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (4) | 1 (4) | 1 (4) | 1 (2)
Neutrophil count decreased (Investigations) | 1 (5) | 0 (0) | 0 (0) | 2 (2)
Platelet count decreased (Investigations) | 1 (10) | 1 (3) | 0 (0) | 3 (5)
White blood cell decreased (Investigations) | 1 (8) | 0 (0) | 1 (4) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (3) | 1 (4) | 1 (2) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5) | 1 (1) | 1 (1) | 2 (3)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 1 (2) | 1 (4) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arterial thromboembolism (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT04714372/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-23): https://cdn.clinicaltrials.gov/large-docs/72/NCT04714372/ICF_001.pdf